CLINICAL TRIAL: NCT05815082
Title: ctDNA-guided Adjuvant Chemotherapy in Liver Metastasis of Colorectal Cancer: A Prospective Multicenter Randomized Controlled Clinical Trial
Brief Title: ctDNA-guided Adjuvant Chemotherapy in Liver Metastasis of Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, Principal Investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1010(CG)2022-02
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer; Liver Metastases; Circulating Tumor Cell; Chemotherapy Effect
Keywords: Colorectal Cancer; Liver Metastases; Circulating Tumor DNA
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watching and waiting group (Experimental): Watch and Wait strategy is one of the treatment strategies of advanced rectal cancer, which recommends no immediate surgery with close surveillance.
  Interventions: Procedure: Colorectal cancer resection combined with liver metastasis resection.
- Adjuvant chemotherapy group (Active Comparator): Chemotherapy regimens recommended include oxaliplatin-based CapeOx or FOLFOX regimens, or single-agent 5-FU/LV, capecitabine, or combination with targeted therapy.
  Interventions: Procedure: Colorectal cancer resection combined with liver metastasis resection.; Drug: FOLFOX chemotherapy regimen

INTERVENTIONS:
Procedure: Colorectal cancer resection combined with liver metastasis resection. — The preferred surgical approach is resection of the corresponding colon segment with regional lymph node dissection. If conditions permit, synchronous resection of the primary lesion and liver metastases of colorectal cancer can be performed to achieve curative resection.
Drug: FOLFOX chemotherapy regimen — Chemotherapy regimens recommended include oxaliplatin-based CapeOx or FOLFOX regimens, or single-agent 5-FU/LV, capecitabine, or combination with targeted therapy.
  Other Names: CapeOx chemotherapy regimen
  Arms: Adjuvant chemotherapy group

SUMMARY:
The goal of this clinical trial is to compare in resectable colorectal cancer liver metastasis patients.The main question it aims to answer is whether the 3-year progression-free survival rate (PFS) of "watching and waiting" is non-inferior to adjuvant chemotherapy in postoperative ctDNA-negative resectable colorectal cancer liver metastasis patients.Participants will undergo ctDNA testing after resection of colorectal cancer liver metastasis, and will be randomly assigned to receive adjuvant chemotherapy or "watching and waiting" treatment strategy. The researchers will compare the outcomes between the two groups to see if the PFS between the two groups is similar.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders are eligible; aged between 18-75 years old; have received neoadjuvant chemotherapy;
2. Patients with liver metastatic colorectal cancer who have achieved R0 resection according to MDT evaluation (including patients with metastases treated with ablation therapy that achieved similar R0 resection effects);
3. Patients with negative ctDNA after surgery;
4. ASA grade <IV and/or ECOG performance status score ≤ 2;
5. Have sufficient understanding of the study and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Patients with distant metastases, including pelvic, ovarian, peritoneal, etc.;
2. Patients with a history of other malignancies;
3. Patients with severe liver, kidney, heart and lung dysfunction, coagulation dysfunction, or serious underlying diseases who cannot tolerate chemotherapy;
4. Patients who are allergic to any component in the study;
5. Patients who have received other tumor-related investigational drug therapy;
6. Patients with severe uncontrolled recurrent infections or other serious uncontrolled concurrent diseases;
7. Patients with other factors that may affect the study results or lead to premature termination of the study, such as alcoholism, drug abuse, other serious diseases that require comprehensive treatment (including mental disorders), and serious abnormal laboratory tests;
8. Patients with a history of severe mental illness;
9. Pregnant or lactating women;
10. Patients with other clinical or laboratory conditions that the investigator deems unsuitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2031-02-20 (Estimated); Study Completion 2033-02-20 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival | 3 years after operation.
  PFS is defined as the time from randomization to the occurrence of any progression or death from any cause.
5-year progression-free survival | 5 years after operation.
  PFS is defined as the time from randomization to the occurrence of any progression or death from any cause.

SECONDARY OUTCOMES:
3-year overall survival | 3 years after operation.
  Overall survival is defined as the time from randomization to death from any cause. For patients who are still alive at the time of the final analysis, the date of the last contact will be recorded.
3-year overall survival | 5 years after operation.
  Overall survival is defined as the time from randomization to death from any cause. For patients who are still alive at the time of the final analysis, the date of the last contact will be recorded.
Complications | 5 years.
  When evaluating the safety and tolerability of adjuvant therapy, researchers typically assess adverse events (AEs) based on their incidence and severity, and then grade them according to the NCI CTCAE version 5.0. NCI CTCAE 5.0 categorizes AEs into 5 grades based on severity, including grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life-threatening), and grade 5 (death).

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliate Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided